CLINICAL TRIAL: NCT00850629
Title: Hormonal Regulation of Body Weight Maintenance
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Charite University, Berlin, Germany (Other)
Collaborators: German Research Foundation (Other)
Responsible Party: Principal Investigator, Professor Joachim Spranger, Professor, Charite University, Berlin, Germany
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: EA2/017/09
Record Dates: First submitted 2009-02-17; First posted 2009-02-25 (Estimated); Last update posted 2018-01-17 (Actual); Status verified 2018-01

CONDITIONS: Obesity; Weight Loss; Weight Gain; Hormone Disturbance; Adipose Tissue; Insulin Resistance; Skeletal Muscle
Keywords: weight regain; endocrine counterregulation
MeSH Terms: conditions — Obesity; Weight Loss; Weight Gain; Endocrine System Diseases; Insulin Resistance

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- placebo (Placebo Comparator): Placebo
  Interventions: Behavioral: placebo
- lifestyle intervention (Experimental): After an initial weight loss, the weight regain will be measured during multimodal lifestyle intervention in children, adolescents and adults
  Interventions: Behavioral: multimodal lifestyle intervention

INTERVENTIONS:
Behavioral: multimodal lifestyle intervention — After an initial weight loss, the weight regain will be measured during multimodal lifestyle intervention in children, adolescents and adults
  Arms: lifestyle intervention
Behavioral: placebo — no intervention, only follow up
  Arms: placebo

SUMMARY:
The investigators here propose to perform a collaborative clinical research effort including a randomized controlled trial investigating the mechanisms of weight maintenance and their relation to a lifestyle intervention in children, adolescents and adults. The detailed investigation and analysis of the variability and dynamics of the endocrine circuits responding to a negative energy balance and weight loss will be accompanied and enhanced by specific clinical projects targeting peripheral and central-nervous aspects of hormonal counter-regulation after weight loss. Mechanisms of endocrine counter-regulation and potential therapeutic approaches will be studied.

ELIGIBILITY:
Inclusion Criteria:

* BMI > 27 kg/m2 (adults)

Exclusion Criteria:

* weight loss of more than 5kg in the last 2 months
* pregnancy, breastfeeding
* patients with:

  * severe heart failure
  * impaired hepatic or renal function
  * anaemia
  * disturbed coagulation (biopsies will not be taken in those subjects)
  * infection, malabsorption
  * severe hypertension
  * cancer within the last 5 years
  * eating disorders or any other psychiatric condition that would interact with the trial intervention
  * any other endocrine disorder
* changes of smoking habits or diets within the last 3 months prior to study inclusion

Ages: 10 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 286 (Actual)
Dates: Start 2010-01 (Actual); Primary Completion 2015-12 (Actual); Study Completion 2016-01 (Actual)

PRIMARY OUTCOMES:
BMI will be assessed during lifestyle intervention in (1) children and adolescents and (2) adults vs. placebo | 21 months
  BMI (kg/m2) will be analyzed after intentional weight loss in two comparable parts of a randomized controlled trial including (1) children and adolescents and (2) adults. Therefore effects of a multimodal lifestyle intervention will be compared to placebo.

SECONDARY OUTCOMES:
Evaluation of leptin during lifestyle intervention | month -3, month 0, month 12, month 18
  Measurement of leptin at baseline, after 3 months of weight loss, as well as after 12 months randomized lifestyle intervention (or placebo) and after additional 6 months follow up
Evaluation of leptin during follow up | 48 months
  Measurement of leptin during follow up until the 48 months
Evaluation of catecholamines during follow up | 48 months
  Measurement of catecholamines during follow up until the 48 months
Evaluation of catecholamines during lifestyle intervention | month -3, month 0, month 12, month 18
  Measurement of catecholamines at baseline, after 3 months of weight loss, as well as after 12 months randomized lifestyle intervention (or placebo) and after additional 6 months follow up
Evaluation of cortisol during lifestyle intervention | month -3, month 0, month 12, month 18
  Measurement of cortisol at baseline, after 3 months of weight loss, as well as after 12 months randomized lifestyle intervention (or placebo) and after additional 6 months follow up
Evaluation of cortisol during follow up | 48 months
  Measurement of cortisol during follow up until the 48 months
Evaluation of glucagon-like peptide 1 (GLP1) during lifestyle intervention | month -3, month 0, month 12, month 18
  Measurement of GLP1 at baseline, after 3 months of weight loss, as well as after 12 months randomized lifestyle intervention (or placebo) and after additional 6 months follow up
Evaluation of GLP1 during follow up | 48 months
  Measurement of GLP1 during follow up until the 48 months
Evaluation of glucose-dependent insulinotropic polypeptide (GIP) during lifestyle intervention | month -3, month 0, month 12, month 18
  Measurement of GIP at baseline, after 3 months of weight loss, as well as after 12 months randomized lifestyle intervention (or placebo) and after additional 6 months follow up
Evaluation of GIP during follow up | 48 months
  Measurement of GIP during follow up until the 48 months
Evaluation of thyroid hormones during lifestyle intervention | month -3, month 0, month 12, month 18
  Measurement of thyroid hormones at baseline, after 3 months of weight loss, as well as after 12 months randomized lifestyle intervention (or placebo) and after additional 6 months follow up
Evaluation of thyroid hormones during follow up | 48 months
  Measurement of thyroid hormones during follow up until the 48 months
Evaluation of insulin during lifestyle intervention | month -3, month 0, month 12, month 18
  Measurement of insulin at baseline, after 3 months of weight loss, as well as after 12 months randomized lifestyle intervention (or placebo) and after additional 6 months follow up
Evaluation of insulin during follow up | 48 months
  Measurement of insulin during follow up until the 48 months
Evaluation of insulin-like growth factor 1 (IGF1) during lifestyle intervention | month -3, month 0, month 12, month 18
  Measurement of IGF1 at baseline, after 3 months of weight loss, as well as after 12 months randomized lifestyle intervention (or placebo) and after additional 6 months follow up
Evaluation of IGF1 during follow up | 48 months
  Measurement of IGF1 during follow up until the 48 months
Evaluation of natriuretic peptide during lifestyle intervention | month -3, month 0, month 12, month 18
  Measurement of natriuretic peptide at baseline, after 3 months of weight loss, as well as after 12 months randomized lifestyle intervention (or placebo) and after additional 6 months follow up
Evaluation of natriuretic peptide during follow up | 48 months
  Measurement of natriuretic peptide during follow up until the 48 months
Evaluation of blood pressure during lifestyle intervention | month -3, month 0, month 12, month 18, month 24, month 36, month 48
  Measurement of blood pressure at baseline, after 3 months of weight loss, as well as after 12 months randomized lifestyle intervention (or placebo) and and after additional 36 months follow up
Evaluation of free fatty acids (FFAs) during lifestyle intervention | month -3, month 0, month 12, month 18, month 24, month 36, month 48
  Measurement of FFAs at baseline, after 3 months of weight loss, as well as after 12 months randomized lifestyle intervention (or placebo) and and after additional 36 months follow up
Evaluation of respiratory coefficient during lifestyle intervention | month -3, month 0, month 12, month 18, month 24, month 36, month 48
  Measurement of respiratory coefficient at baseline, after 3 months of weight loss, as well as after 12 months randomized lifestyle intervention (or placebo) and and after additional 36 months follow up
Measurement of messenger ribonucleic acid (mRNA) changes in adipose and skeletal muscle before (T-3), after weight loss (T0) and after as well as after 12 months randomized lifestyle intervention (or placebo) | month -3, month 0, month 12
  Measurement of systemic and tissue specific changes in adipose tissue and skeletal muscle using RNA sequencing (counts)
Measurement of insulin sensitivity | month -3, month 0, month 12
  Measurement of systemic and tissue specific changes in adipose and muscle insulin sensitivity using hyperinsulinemic clamp (mg•kg-1•min-1/(mU•L-1)) before (T-3), after weight loss (T0) and after as well as after 12 months randomized lifestyle intervention (or placebo)
Prediction of body weight regain | month 18, month 48
  No additional measurement will be done. However, we will analyse the predictive impact of already measured parameters on long-term course of BMI (18 and 48 months) using mathematical models
Prediction of insulin sensitivity | month 18, month 48
  No additional measurement will be done. However, we will analyse the predictive impact of already measured parameters on insulin sensitivity (18 and 48 months) using mathematical models
Prediction of energy expenditure | month 18, month 48
  No additional measurement will be done. However, we will analyse the predictive impact of already measured parameters on energy expenditure (18 and 48 months) using mathematical models
Prediction of muscle mass | month 18, month 48
  No additional measurement will be done. However, we will analyse the predictive impact of already measured parameters on muscle mass (18 and 48 months) using mathematical models
Prediction of fat mass | month 18, month 48
  No additional measurement will be done. However, we will analyse the predictive impact of already measured parameters on fat mass (18 and 48 months) using mathematical models
BMI course after a lifestyle intervention in (1) children and adolescents and (2) adults vs. placebo | month 24, month 36, month 48
  BMI (kg/m2) after the randomized control trial (RCT) (18 months) will be analyzed up to 48 months.
changes of fatty acids during the intervention | month -3, month 0, month 12, month 18, month 24, month 36, month 48
  Analysis of fatty acids at baseline, after 3 months of weight loss, as well as after 12 months randomized lifestyle intervention (or placebo) and and after additional 36 months follow up
changes acylcarnitines | month -3, month 0
  Analysis of acylcarnitines at baseline and after 3 months of weight loss
changes acylcarnitines | month 12, month 18, month 24, month 36, month 48
  Analysis of acylcarnitines after 12 months randomized lifestyle intervention (or placebo) and and after additional 36 months follow up
body composition | month -3, month 0, month 12, month 18, month 24, month 36, month 48
  Whole body fat mass (kg, %) will be measured at baseline, after 3 months of weight loss, as well as after 12 months randomized lifestyle intervention (or placebo) and and after additional 36 months follow up

CONTACTS AND LOCATIONS:
Overall Officials: Knut Mai, Prof, Principal Investigator — Charite
Locations (1):
- Charite, Berlin, Germany

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Haberbosch L, Kierszniowska S, Willmitzer L, Mai K, Spranger J, Maurer L. 5-Aminovaleric acid betaine predicts impaired glucose metabolism and diabetes. Nutr Diabetes. 2023 Sep 20;13(1):17. doi: 10.1038/s41387-023-00245-3. PMID 37730732
- [Derived] Li L, Soll D, Leupelt V, Spranger J, Mai K. Weight loss-induced improvement of body weight and insulin sensitivity is not amplified by a subsequent 12-month weight maintenance intervention but is predicted by adaption of adipose atrial natriuretic peptide system: 48-month results of a randomized controlled trial. BMC Med. 2022 Jul 28;20(1):238. doi: 10.1186/s12916-022-02435-9. PMID 35897098
- [Derived] Soll D, Gawron J, Pletsch-Borba L, Spranger J, Mai K. Long-term impact of the metabolic status on weight loss-induced health benefits. Nutr Metab (Lond). 2022 Mar 28;19(1):25. doi: 10.1186/s12986-022-00660-w. PMID 35346256
- [Derived] Li L, Spranger L, Stobaus N, Beer F, Decker AM, Wernicke C, Brachs S, Brachs M, Spranger J, Mai K. Fetuin-B, a potential link of liver-adipose tissue cross talk during diet-induced weight loss-weight maintenance. Nutr Diabetes. 2021 Oct 5;11(1):31. doi: 10.1038/s41387-021-00174-z. PMID 34611132
- [Derived] Li L, Spranger L, Soll D, Beer F, Brachs M, Spranger J, Mai K. Metabolic impact of weight loss induced reduction of adipose ACE-2 - Potential implication in COVID-19 infections? Metabolism. 2020 Dec;113:154401. doi: 10.1016/j.metabol.2020.154401. Epub 2020 Oct 13. PMID 33065163
- [Derived] Brachs S, Polack J, Brachs M, Jahn-Hofmann K, Elvert R, Pfenninger A, Barenz F, Margerie D, Mai K, Spranger J, Kannt A. Genetic Nicotinamide N-Methyltransferase (Nnmt) Deficiency in Male Mice Improves Insulin Sensitivity in Diet-Induced Obesity but Does Not Affect Glucose Tolerance. Diabetes. 2019 Mar;68(3):527-542. doi: 10.2337/db18-0780. Epub 2018 Dec 14. PMID 30552109
- [Derived] Mai K, Li L, Wiegand S, Brachs M, Leupelt V, Ernert A, Kuhnen P, Hubner N, Robinson P, Chen W, Krude H, Spranger J. An Integrated Understanding of the Molecular Mechanisms of How Adipose Tissue Metabolism Affects Long-term Body Weight Maintenance. Diabetes. 2019 Jan;68(1):57-65. doi: 10.2337/db18-0440. Epub 2018 Nov 2. PMID 30389745
- [Derived] Bau AM, Ernert A, Krude H, Wiegand S. Hormonal regulatory mechanisms in obese children and adolescents after previous weight reduction with a lifestyle intervention: maintain - paediatric part - a RCT from 2009-15. BMC Obes. 2016 Jun 10;3:29. doi: 10.1186/s40608-016-0110-8. eCollection 2016. PMID 27298729
- [Derived] Brachs M, Wiegand S, Leupelt V, Ernert A, Kintscher U, Jumpertz von Schwarzenberg R, Decker AM, Bobbert T, Hubner N, Chen W, Krude H, Spranger J, Mai K. ANP system activity predicts variability of fat mass reduction and insulin sensitivity during weight loss. Metabolism. 2016 Jun;65(6):935-43. doi: 10.1016/j.metabol.2016.03.013. Epub 2016 Apr 7. PMID 27173472
- [Derived] Weygandt M, Mai K, Dommes E, Ritter K, Leupelt V, Spranger J, Haynes JD. Impulse control in the dorsolateral prefrontal cortex counteracts post-diet weight regain in obesity. Neuroimage. 2015 Apr 1;109:318-27. doi: 10.1016/j.neuroimage.2014.12.073. Epub 2015 Jan 7. PMID 25576647